CLINICAL TRIAL: NCT03692247
Title: Quantitative Sensory Testing in Response to Music Interventions
Brief Title: The Impact of Music Therapy on Nociceptive Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Edward W Boyer, Director of Academic Development, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017P002872
Record Dates: First submitted 2018-06-16; First posted 2018-10-02 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Pain; Chronic Pain
Keywords: pain; music
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: This is a cohort study of one group of 60 healthy volunteers without a diagnosis of neuropathy or chronic pain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quantitative Sensory Testing (Other): After answering brief questionnaires assessing psychosocial factors related to anxiety, catastrophizing, and pain, participants will undergo quantitative sensory tests where they will use a simple numeric rating scale (0-10) to rate pain and anxiety at several points during two QST sessions. During the second QST session, participants will use Unwind, a smartphone-based music intervention.
  Interventions: Other: Smartphone-based Music Intervention

INTERVENTIONS:
Other: Smartphone-based Music Intervention — The smartphone-based music intervention (Unwind) is a music protocol that gathers basic information from the patient including a 0-10 pain scale and 0-10 anxiety scale as well as recorded heart rate. Using these variables, a machine learning protocol pieces together a music intervention between 5-20 minutes long. The duration of the intervention can be controlled by the patient or experimenter. No identifying data is kept on the smartphone.

SUMMARY:
The purpose of this study is to understand the use of brief, personalized music interventions to decrease pain. Persisting and recurring pain is devastating to individuals and society. The worry and anxiety people feel while experiencing chronic pain may increase how much pain they feel. Enjoyable music feels good and affects brain chemicals in a way that can lessen feelings of pain. Music that feels good can also lower the anxiety and worry that accompany chronic pain which may play a role in the pain relief music provides.

DETAILED DESCRIPTION:
Chronic pain is devastating to individuals and society. Individuals who experience chronic pain have poorer health outcomes, utilize increased healthcare resources and have higher rates of disability. At present, treatment of chronic pain is limited to behavioral interventions and pharmacologic interventions. Many individuals with chronic pain will use opioid analgesics at some point in the continuum of pain. Prolonged use of opioid analgesics--even for durations as short as 3 days puts individuals at risk for nonmedical opioid use, addiction, and may fuel transitions from oral opioids to heroin.

Outside of the original insult precipitating chronic pain, increasing evidence suggests that individual factors such as anxiety and catastrophizing are associated with development of chronic pain and increased painful response to stimuli. It is therefore suggestive that treating underlying causes of anxiety and catastrophizing may lead to novel adjunctive therapies to manage chronic pain.

Music is emotive and known to modulate affect. Music that "feels good" has been described to modulate the dopaminergic and serotonin reward pathways in the brain thereby improving positive affect. Improved affect counteracts negatively valenced affect like depression, anxiety, and catastrophizing, and may be able to modulate the individual response to pain. The purpose of this pilot study is to investigate the acceptability and feasibility of a smartphone-based app on healthy volunteers.

In order to measure the impact of the music app on individual responses to pain, the investigators will use quantitative sensory testing (QST) to induce a mild-moderate, standardized pain stimulus, and measure participants' pain in the absence and presence of this music intervention. The QST is a 10 minute session that includes a set of sensory tests, which elicit a mild to moderate painful response, including a pressure pain threshold and tolerance using a handheld digital algometer, the temporal summation of pain using a set of weighted pinprick probes, and immersing hand in cold water. Primary outcome will be the modulation of pain scores by music, and secondary outcomes will include the impact of music on anxiety and catastrophizing, using brief, validated questionnaires, and whether changes in these measures of affect mediate any impact on pain processing.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Able to sign English written consent
* No history of chronic opioid use (have an opioid prescription more than 30 days).

Exclusion Criteria:

* Under 18 years old
* Non-English speaking
* Unwilling to undergo quantitative sensory testing
* Hearing loss
* Diagnosis of neuropathy
* History of chronic opioid use (having an opioid prescription more than 30 days).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Sensitivity in the Presence of Music | 40 minutes
  Change in pain sensitivity, measured as a difference in the temporal summation of pain with a mechanical stimulus between a control and music condition of testing.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Boyer, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No